CLINICAL TRIAL: NCT02938663
Title: Cultural Factors Underlying Obesity in African-American Adolescents
Brief Title: Health & Culture Project: Cultural Factors Underlying Obesity in African-American Adolescents
Acronym: HCP
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Rebecca Hasson, Director, Childhood Disparities Research Laboratory, University of Michigan
Other Study IDs: HUM00080820
Record Dates: First submitted 2016-10-01; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Surveys and Questionnaires; Weights and Measures

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionnaires and measurements: assessment of physical activity, dietary intake, psychosocial factors, weight status
  Interventions: Behavioral: Questionnaires and Measurements

INTERVENTIONS:
Behavioral: Questionnaires and Measurements — Participants completed anthropometric measurements and questionnaires assessing psychosocial stress, habitual dietary intake and physical activity as well as cultural identity, identity-based motivation and socioeconomic status. At home, participants recorded their habitual physical activity and food intake. Participants then returned to the laboratory to complete an assessment of identity-based motivation and received personalized information regarding their habitual physical activity and dietary patterns.

SUMMARY:
The overall goal of this study is to examine the relationships between cultural identity and identity-based motivation, physical activity, diet and obesity risk in African-American adolescents. It was hypothesized that African-American youth who self-report a bicultural identity maintain health promotion beliefs and behaviors that reduce obesity risk compared to minority youth who only identify with one culture or neither culture. It was also hypothesized that African-American youth who self report a bicultural identity are more likely to hold beliefs about health promotion behaviors that are congruent with their cultural identity than compared to youth who only identify with one culture or neither culture.

DETAILED DESCRIPTION:
Obesity is a significant problem in African-American adolescents in the United States (US). The most recent data suggests a doubling of overweight (BMI percentile > 85th for age and gender) and obesity (BMI percentile >95th for age and gender) among these racial/ethnic minority youth in the last 10 years. In 2007-8, 39.5% of African-Americans a ages 12-19 were overweight and 24.4% were obese. These obesity rates were approximately double that of non-Latino whites. Until now, most of our efforts to reduce pediatric obesity have targeted at-risk youth who are physically inactive and over-consume energy dense foods. More recently, however, that focus has broadened as a result of new understanding about how cultural factors also shape physical activity behaviors and dietary patterns. With the rapid increase in cultural diversity of the US, Black culture is quickly becoming a part of mainstream American culture, evolving within the US, while simultaneously integrating aspects of different African and Black American cultures. Consequently, African- American youth who come of age in the US, a multicultural society, interact with people from different cultural backgrounds that can lead to an interchange of cultural attitudes, beliefs and behaviors. Specifically, these youth may adopt one of four general cultural identities: (a) bicultural identity-combining aspects of their family's culture with aspects of mainstream American culture; (b) US cultural identity- replacing their family's culture with mainstream American culture; (c) traditional cultural identity- retaining their family's culture while rejecting mainstream American culture; or (d) marginalized cultural identity- becoming alienated from both cultures. Biculturalism is considered the most adaptive process allowing individuals to function effectively in a multicultural society while still maintaining supportive connections to their own family's culture. Hence, it was hypothesized that racial/ethnic minority youth who self-report a bicultural identity maintain health promotion beliefs and behaviors that reduce obesity risk compared to minority youth who only identify with one culture or neither culture.

Empirical investigations assessing the impact of cultural identity on health promotion behaviors in African-American adults have reported a positive identification with African-American culture and a self- perception of being successful in both the "black" and "white" ways of life were associated with health promotion behaviors including reduced fat consumption and more participation in leisure-time physical activity. Less is known about the impact of cultural identity on physical activity behavior and dietary patterns in African-American youth. One important mechanism underlying the link between cultural identity, physical activity and diet likely involves identity-based motivation the process by which individuals see health behaviors as being congruent or incongruent with their cultural identity. According to the identity-based motivation model, health promotion behaviors (e.g., exercising, restraining eating, reducing fat and sugar intake) are not simply personal choices made in the moment but rather are identity-infused habits. Hence, ethnic minorities who view health promotion behaviors as White and middle-class and unhealthy behaviors (e.g., high-fat, high-sugar diet, sedentary behaviors) as a defining characteristic of their own cultural identity are less likely to engage in health promotion behaviors. Oyserman et al argues that even though physical activity and diet have important consequences for health, these identity-infused behaviors are engaged in less for their health consequences than for their identity consequences. Hence, identity-based motivation may serve as a novel mechanism explaining the link between cultural identity, physical activity and diet, ultimately influencing obesity risk in African-American youth. It was hypothesized that racial/ethnic minority youth who self report a bicultural identity are more likely to hold beliefs about health promotion behaviors that are congruent with their cultural identity than compared to youth who only identify with one culture or neither culture.

1. Test whether a bicultural identity among African-American adolescents is associated with obesity risk and related health behaviors.

   H1: African-American adolescents who self-report a bicultural identity will report lower BMIs, increased physical activity and lower fat and sugar intake compared to adolescents who maintain an alternate cultural identity.
2. Test whether a bicultural identity is associated with identity-based motivation in African-American adolescents.

   H2: African-American adolescents who self-report a bicultural identity view health promotion behaviors as identity-congruent compared to adolescents who maintain an alternate cultural identity.
3. To evaluate whether identity-based motivation mediates the associations between a bicultural identity, obesity risk and related health behaviors in African-American adolescents. H3: Identity-congruent health promotion beliefs mediate associations between biculturalism, BMI, physical activity and diet in African-American adolescents.

The Health & Culture project represents the convergence of two rapidly expanding areas of pediatric obesity research; the role of cultural identity and identity-based motivation in shaping health promotion behaviors. The investigators recently submitted several papers for publication examining associations between cultural identity, physical activity, diet and diabetes-related metabolic risk factors in obese African- American adolescents. Results demonstrate that for obese African-American adolescents, biculturalism was negatively associated with diabetes risk (via increased pancreatic beta-cell function assessed during a frequently-sampled intravenous glucose tolerance test). These relationships remained significant after controlling for household socioeconomic status, sex, pubertal maturation, fat/fat-free mass, physical activity and diet. These exciting findings peeked our interest in the area of cultural psychology, particularly as it relates to racial/ethnic disparities in pediatric obesity. Moreover, these preliminary data extend the findings of others who have pointed to the important role of cultural identity in shaping health and health behaviors. The researchers are advancing this area of research further by examining the influence of identity-based motivation in the context of cultural identity. Because identity-based motivation is a modifiable psychosocial mechanism, a richer and more in depth understanding of how identity-based motivation may help to inform culturally-tailored interventions could have a large public health impact by improving health promotion behaviors in racial/ethnic minority youth and reducing the economic burden of pediatric obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 12-18 years old from the greater Ann Arbor and Ypsilanti, Michigan areas were recruited to participate in this study.

Exclusion Criteria:

Adolescents were not be eligible for the study if any of the following apply:

* Participated in a weight loss or exercise program within the previous 6 months;
* Were taking any medications known to influence body composition;
* Diagnosed with syndromes or diseases that may influence body composition and fat distribution;
* Previously diagnosed with any major illness/health condition since birth.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: African American children and adolescents were recruited to participate in this study. The study included both genders aged 12-18 years. Adolescents were chosen because pubertal youth are at increased risk for obesity than pre-pubertal children.
Sampling Method: Non-Probability Sample
Enrollment: 273 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
body mass index | 1 day
  Weight and height were measured to the nearest 0.1 kg and 0.1 cm, respectively, using a beam medical scale and wall-mounted stadiometer. BMI and BMI percentiles were determined.

SECONDARY OUTCOMES:
Dietary intake | 3 days
  Participants recorded their daily food intake for 3 days using dietary food records.
Cultural Identity | 1 day
  Participants completed the Acculturation, Habits, and Interests Multicultural Scale for Adolescents.
Identity-based motivation | 1 day
  Participants completed the Identity-based motivation questionnaire.
Minutes of moderate-to-vigorous physical activity | 7-14 days
  Participants wore an accelerometer for 7-14 days at home. Moderate-to-vigorous physical activity was calculated from accelerometer data.
Dietary fat intake attitudes and beliefs | 1 day
  Participants completed the Physician-based Assessment & Counseling for Exercise (PACE) Adolescent dietary questionnaire to assess their attitudes and beliefs regarding dietary fat intake.
Fruit and vegetable attitudes and beliefs | 1 day
  Participants completed the Physician-based Assessment & Counseling for Exercise (PACE) Adolescent dietary questionnaire to assess their attitudes and beliefs regarding fruit and vegetable intake.
Eating Attitudes | 1 day
  Participants completed the eating attitudes to assess their beliefs and attitudes about food.
Physical activity attitudes and beliefs | 1 day
  Participants completed the Physician-based Assessment & Counseling for Exercise (PACE) Adolescent questionnaire to assess their attitudes and beliefs regarding physical activity participation.
Sedentary behaviors attitudes and beliefs | 1 day
  Participants completed the Physician-based Assessment & Counseling for Exercise (PACE) Adolescent questionnaire to assess their attitudes and beliefs regarding sedentary behaviors
Exposure to discrimination | 1 day
  Participants completed the Adolescent Discrimination Distress Index to assess their exposure and perceived impact of racial discrimination in their lives
Parental stress | 1 day
  Parents of participants answered the CRYSIS questionnaire to assess parental stress levels
Acute daily stress | 1 day
  Participants completed the Daily stress inventory to assess their exposure to daily acute stressors.
Parent perceptions of their child's health environment | 1 day
  Parent's of participants answer the Physician-based Assessment & Counseling for Exercise (PACE) Health and environment survey to assess their perceptions of their child's access to health resources in the home and community environment.
Lifestyle choices | 1 day
  Participants completed the Lifestyle questionnaire assessing their lifestyle choices (e.g. wearing seat belts, getting 8 hours of sleep, etc).
Perceived social status | 1 day
  Participants completed the MacArthur Scale of Subjective Social Status- Youth Version Questionnaire to assess their perceived status within their school and community.
Household demographics | 1 day
  Parent's of participants answered the Parent questionnaire to quantify household characteristics.
Perceived chronic stress | 1 day
  Participants answered the Perceived Stress Scale to assess their levels of perceived stress.
Pubertal development | 1 day
  Participants answered the Pubertal development scale to assess their level of pubertal development
Stress coping | 1 day
  Participants answered the Schoolager's Coping Strategies Inventory to assess ways in which they cope with their stress.
Self-esteem | 1 day
  Participants answered completed the Sorenson Self-Esteem Test to assess their level of self-esteem.
Exposure to community violence | 1 day
  Participants answered the Survey of Children's exposure to community violence to assess their exposure to community violence.
Dietary intake | 1 day
  Participants completed the food frequency questionnaire to assess their dietary intake over the past year.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca E Hasson, Principal Investigator — University of Michigan
Locations (1):
- Childhood Disparities Research Laboratory, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ajibewa TA, Robinson LE, Toledo-Corral C, Miller AL, Sonneville KR, Hasson RE. Acute Daily Stress, Daily Food Consumption, and the Moderating Effect of Disordered Eating among Adolescents with Overweight/Obesity. Child Obes. 2021 Sep;17(6):391-399. doi: 10.1089/chi.2021.0017. Epub 2021 Apr 26. PMID 33902320
- [Derived] Ajibewa TA, Beemer LR, Sonneville KR, Miller AL, Toledo-Corral C, Robinson LE, Hasson RE. Psychological Stress and Lowered Physical Activity Enjoyment in Adolescents With Overweight/Obesity. Am J Health Promot. 2021 Jul;35(6):766-774. doi: 10.1177/0890117121997042. Epub 2021 Feb 25. PMID 33626891
- [Derived] Allport L, Song M, Leung CW, McGlumphy KC, Hasson RE. Influence of Parent Stressors on Adolescent Obesity in African American Youth. J Obes. 2019 Dec 1;2019:1316765. doi: 10.1155/2019/1316765. eCollection 2019. PMID 31871784
- [Derived] Nagy MR, McGlumphy KC, Dopp R, Lewis TC, Hasson RE. Association between asthma, obesity, and health behaviors in African American youth. J Asthma. 2020 Apr;57(4):410-420. doi: 10.1080/02770903.2019.1571083. Epub 2019 Jan 31. PMID 30702005
- [Derived] Shaver ER, McGlumphy KC, Gill AK, Hasson RE. Application of the Transtheoretical Model to Physical Activity and Exercise Behaviors in African-American Adolescents. Am J Health Behav. 2019 Jan 1;43(1):119-132. doi: 10.5993/AJHB.43.1.10. PMID 30522571
- [Derived] McGlumphy KC, Shaver ER, Ajibewa TA, Hasson RE. Perceived Stress Predicts Lower Physical Activity in African-American Boys, but not Girls. Am J Health Behav. 2018 Mar 1;42(2):93-105. doi: 10.5993/AJHB.42.2.9. PMID 29458518
- [Derived] Nelson DS, Gerras JM, McGlumphy KC, Shaver ER, Gill AK, Kanneganti K, Ajibewa TA, Hasson RE. Racial Discrimination and Low Household Education Predict Higher Body Mass Index in African American Youth. Child Obes. 2018 Feb/Mar;14(2):114-121. doi: 10.1089/chi.2017.0218. Epub 2017 Dec 6. PMID 29211516